CLINICAL TRIAL: NCT01780714
Title: A Single-center, Open-label, Randomized, Controlled, 2-arm Parallel Group Study to Evaluate the Exposure to Selected Smoke Constituents in Smoking, But Otherwise Healthy Subjects Switching From Conventional Cigarettes to the Tobacco Heating System (THS) 2.1
Brief Title: Exploratory THS 2.1 Biomarkers of Exposure Study
Acronym: ZRHX-EX-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZRHX-EX-01
Record Dates: First submitted 2013-01-15; First posted 2013-01-31 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Smoking
Keywords: smoking; cigarette; exposure; biomarker; human smoking topography (HST); modified risk tobacco product (MRTP); THS 2.1
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional cigarettes (CC) (Active Comparator): Smokers are continuing to smoke exclusively their usual own brand of CC, for 5 days, ad libitum, under highly controlled conditions
  Interventions: Other: Conventional cigarettes (CC)
- Tobacco Heating System 2.1 (THS 2.1) (Experimental): Smokers are switching to the exclusive and ad-libitum use of THS 2.1 for 5 days, under highly controlled conditions
  Interventions: Other: THS 2.1

INTERVENTIONS:
Other: Conventional cigarettes (CC) — Subjects are randomized in a 1:1 fashion to be assigned either A) continuing CC, or B) switching to THS 2.1
  Arms: Conventional cigarettes (CC)
Other: THS 2.1 — Subjects are randomized in a 1:1 fashion to be assigned either A) continuing CC, or B) switching to THS 2.1
  Arms: Tobacco Heating System 2.1 (THS 2.1)

SUMMARY:
The goal of this exploratory study is to evaluate the effect of a candidate modified risk tobacco product (MRTP), THS 2.1, on selected biomarkers of exposure to harmful and potentially harmful smoke constituents (HPHCs), compared to conventional cigarettes (CC). The subjective effects (urge to smoke and withdrawal symptoms) which are related to the use of this product will be explored. Initial information on safety and on some biological effects when using THS 2.1 will be collected. Human Smoking Topography (HST) will be explored.

DETAILED DESCRIPTION:
This study intends to evaluate the levels of selected biomarkers of exposure to selected HPHC and of cytochrome P450 1A2 (CYP1A2) enzymatic activity, as compared to smokers continuing smoking CC ad libitum, after 5 days of ad libitum use.

Additional parameters will be explored, such as: cytochrome P450 2A6 (CYP2A6) enzymatic activity, nicotine pharmacokinetics, product evaluation and safety, marker of platelet function, and HST.

After screening, subjects will be admitted to the clinic for 9 days, including the Day of Admission, 2 days of baseline during which all subjects will continue to smoke their usual CC for a 5-day exposure after randomization. After leaving the clinic on the Day of Discharge, the subjects will be followed up for safety over a period of 7 days. All subjects will receive smoking cessation advice at screening, at Day of Admission and at Day of Discharge.

This clinical study will be conducted in compliance with International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use (ICH Good Clinical Practice), the Declaration of Helsinki as amended in 2008, and the applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed an informed consent form before commencement of study procedures
* Healthy Caucasian aged between 23 to 65 years
* Subject is a current smoker for at least 3 years (based on self-reporting and biochemically verified), who, for the last 4 weeks, had smoked at least 10 commercially available non-mentholated CC per day, and is not planning to make a quit attempt within the next 3 months

Main Exclusion Criteria:

* As per Investigator judgment, the subject should not participate in the study for any reason (e.g. medical, psychiatric and/or social reason)
* The subject has a medical condition requiring smoking cessation, or has a clinically relevant disease / condition which could interfere with the study participation and/or study results
* The subject has participated in a clinical study within 3 months prior to the Screening Visit
* Pregnant or lactating woman, and for woman of childbearing potential, absence / refusal to use an acceptable method of effective contraception

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of carboxyhemoglobin (COHb) levels in blood, and evaluation of excretion of 3-hydroxypropyl mercapturic acid (3-HPMA), monohydroxybutenyl mercapturic acid (MHBMA), and S-phenyl mercapturic acid (S-PMA) in 24-hour urine on switching to THS 2.1 | 5 days
  Biomarkers of exposure to carbon monoxide (CO), acrolein, 1,3-butadiene, and benzene

SECONDARY OUTCOMES:
Selected secondary biomarkers of exposure to HPHCs | 5 days
  Evaluation of the levels of total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (total NNAL),1-hydroxypyrene , total N-nitrosonornicotine (NNN), 4-aminobiphenyl (4-ABP), 2- aminonaphthalene (2-NA), o-toluidine, nicotine equivalents and 2-cyanoethylmercapturic acid, biomarkers of exposure to the HPHCs 4-(methylnitrosamino)-1- (3-pyridyl)-1-butanone, NNN, 4-ABP, 2-NA, o-toluidine, nicotine and acrylonitrile, respectively, as excreted in urine.
CYP1A2 activity and CYP2A6 activity | 5 days
  Evaluation of the CYP1A2 activity, as measured by the plasma caffeine molar metabolic ratio (paraxanthine / caffeine) and in CYP2A6 activity, as measured by nicotine molar metabolic ratio (3-hydroxy-cotinine / cotinine) in plasma and in urine
Plasma nicotine | 5 days
  Time course of nicotine plasma concentrations and derived pharmacokinetic parameters
11-dehydro-thromboxane B2 (11-DTX-B2) | 5 days
  To describe the 11-DTX-B2 levels in urine as a marker of platelet function
Product use and smoking topography | Up to 5 days
  Monitoring of daily product use and human smoking topography
Safety monitoring | 8 days + 7 days follow-up
  Monitoring of adverse events, based on clinical and laboratory evaluation
Cough Visual Analog Scale (Cough VAS) | 7 days
  Visual Analog Scale on cough
Modified Cigarette Evaluation Questionnaire (MCEQ) | 5 days
  MCEQ measuring subjective effects of smoking
Questionnaire on Smoking Urges (brief version) (QSU-brief) | 5 days
  QSU-brief measuring subjective effects of smoking
Minnesota Withdrawal Scale-Revised (MNSWS-R) | 5 days
  MNWS-R questionnaire measuring subjective effects of smoking

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Jarus-Dziedzic, MD PhD, Principal Investigator — MTZ Clinical Research Sp. z o.o., Warsaw, Poland
Locations (1):
- MTZ Clinical Research Sp. z o.o., Warsaw, Poland

REFERENCES:
- [Result] Ludicke F, Baker G, Magnette J, Picavet P, Weitkunat R. Reduced Exposure to Harmful and Potentially Harmful Smoke Constituents With the Tobacco Heating System 2.1. Nicotine Tob Res. 2017 Feb;19(2):168-175. doi: 10.1093/ntr/ntw164. Epub 2016 Jul 1. PMID 27613951